CLINICAL TRIAL: NCT03867669
Title: Neurodevelopmental Outcomes at Three Years of Age in Very Preterm Infants (< 31 Weeks Gestational Age) or Very Low Birth Weight (< 1500 Grams) Randomized to Single Patient Rooms Compared to Open Bay Neonatal Intensive Care Unit
Brief Title: Single Patient Room Versus Open Bay in NICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Principal Investigator, Mike Vincer, Michael Vincer, Staff Neonatologist, Medical Director Perinatal Follow Up Program, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Single room vs open bay
Record Dates: First submitted 2018-10-31; First posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Neurodevelopmental Outcomes
Keywords: Developmental Disabilities; Follow-Up Studies; Infant, Premature; Intensive Care Units, Neonatal; randomized controlled trial
MeSH Terms: conditions — Developmental Disabilities; Premature Birth | interventions — Patients' Rooms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Patient Room (Experimental): Patients randomized to this arm will be admitted to a NICU single patient room.
  Interventions: Other: Single patient room
- Open Bay (Placebo Comparator): Patients randomized to this arm will be admitted to the open bay NICU Unit.
  Interventions: Other: Open Bay Unit

INTERVENTIONS:
Other: Open Bay Unit — The eligible infants will be randomized at birth/admission to either the single patient room (experimental) or the open bay unit (Comparator)
  Arms: Open Bay
Other: Single patient room — The eligible infants will be randomized at birth/admission to either the single patient room (experimental) or the open bay unit (Comparator)
  Arms: Single Patient Room

SUMMARY:
The NICU at the IWK Health Center in Halifax, Nova Scotia is embarking on a redevelopment project that will see its current open bay design converted to a single room care environment. There will be a period during the redevelopment when new single room care unit will coexist with one open bay unit. This provides a unique opportunity to explore the effect of the two different environmental designs on both short and long-term outcomes. Preterm infants (under 31 weeks gestational age) and very low birth weight infants (under 1500 grams) will be randomized to either the open bay unit or the single patient room unit, at 36 months corrected age neurodevelopmental outcomes will be assessed.

DETAILED DESCRIPTION:
Do very preterm infants (< 31 weeks gestational age) and very low birth weight infants (< 1500 grams) admitted to a single patient room in the NICU have improved long-term neurodevelopmental outcomes when compared to very preterm infants admitted to an open bay in the NICU?

Babies who will be admitted to NICU will be randomized to either the open-bay unit or single room care. The randomization will be achieved through the use of the WANNNT (Winnipeg Assessment of Neonatal Nurses Need Tool) and current patient census; this involves taking 1/3 of the fraction of the patient census on each team and adding it to 2/3 of the fraction of the WANNNT. This methodology was reviewed by several IWK Committees including Ethics, Family Leadership Council, Neonatal care Committee and the Family Centered Care Committee. This randomization is designed to ensure fairness and an equitable workload between the two units.

Eligible study infants are also enrolled in the Perinatal Follow-Up Program (PFU) as a standard of care at the IWK Health Center. The baby's legal guardian signs a consent to be enrolled in the PFU Program and to allow collection and use of data for their child as long as their child cannot be identified from the use of the data. All families of infants admitted to NICU, whether or not they have been enrolled in the PFU Program will receive an information package explaining the single patient room NICU compared with the open bay NICU.

At three years of corrected gestational age, all eligible infants will have the Bayley Scales of Infant and Toddler Development - version 3 assessment completed which evaluates cognitive, language and motor skills. These infants will also be examined for the presence or absence of cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* All very preterm infants born less than 31 weeks gestational age or birth weight less than or equal to 1500 grams
* age less than 14 days
* Multiples will be randomized to the same arm.

Exclusion Criteria:

* Babies with major anomalies
* Babies admitted for palliative care only

Max Age: 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with neurodevelopmental impairment or death | From randomization to age 36 months corrected age
  adverse neurodevelopmental outcome including any of the following: 1. Cerebral palsy, 2. Bayley-III scores (cognitive or language <85), 3. Blindness (vision <20/200 in the best eye) 4. Deafness (bilateral) requiring hearing aids for correction; or 5. Death prior to 36 months corrected gestational age.

SECONDARY OUTCOMES:
Number of Participants with cerebral palsy | From randomization to age 36 months corrected age
  any degree of cerebral palsy (minor = level 1 or 2) (major = level 3-5)
Number of participants who died | From randomization to age 36 months corrected age
  Death before 36 months corrected age
Number of Participants with low cognitive scores (<85) of the Bayley Scales of Infant and Toddler Development (version III) | From randomization to age 36 months corrected age
  <85 on the Bayley Scales of Infant and Toddler Development (version III) represents -1 standard deviations below the mean. (Scale range is 55-145, higher scores are better)
Number of Participants with low language scores (<85) of the Bayley Scales of Infant and Toddler Development (version III) | From randomization to age 36 months corrected age
  <85 on the Bayley Scales of Infant and Toddler Development (version III) which represents -1 standard deviations below the mean. (Scale range is 45-155, higher scores are better)
Number of Participants with low motor scores (<85) of the Bayley Scales of Infant and Toddler Development (version III) | From randomization to age 36 months corrected age
  <85 on the Bayley Scales of Infant and Toddler Development (version III) which represents -1 standard deviations below the mean. (Scale range is 45-155, higher scores are better)
Number of participants with blindness | From randomization to age 36 months corrected age
  vision <20/200 in the best eye
Number of participants with deafness | From randomization to age 36 months corrected age
  Deafness (bilateral) requiring hearing aids for correction

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vincer, Principal Investigator — Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domanico R, Davis DK, Coleman F, Davis BO. Documenting the NICU design dilemma: comparative patient progress in open-ward and single family room units. J Perinatol. 2011 Apr;31(4):281-8. doi: 10.1038/jp.2010.120. Epub 2010 Nov 11. PMID 21072040
- [Background] Erdeve O, Arsan S, Canpolat FE, Ertem IO, Karagol BS, Atasay B, Yurdakok M, Tekinalp G, Turmen T. Does individual room implemented family-centered care contribute to mother-infant interaction in preterm deliveries necessitating neonatal intensive care unit hospitalization? Am J Perinatol. 2009 Feb;26(2):159-64. doi: 10.1055/s-0028-1095186. Epub 2008 Nov 19. PMID 19021100
- [Background] Lester BM, Hawes K, Abar B, Sullivan M, Miller R, Bigsby R, Laptook A, Salisbury A, Taub M, Lagasse LL, Padbury JF. Single-family room care and neurobehavioral and medical outcomes in preterm infants. Pediatrics. 2014 Oct;134(4):754-60. doi: 10.1542/peds.2013-4252. Epub 2014 Sep 22. PMID 25246623
- [Background] Lester BM, Salisbury AL, Hawes K, Dansereau LM, Bigsby R, Laptook A, Taub M, Lagasse LL, Vohr BR, Padbury JF. 18-Month Follow-Up of Infants Cared for in a Single-Family Room Neonatal Intensive Care Unit. J Pediatr. 2016 Oct;177:84-89. doi: 10.1016/j.jpeds.2016.06.069. Epub 2016 Jul 26. PMID 27470693
- [Background] Ortenstrand A, Westrup B, Brostrom EB, Sarman I, Akerstrom S, Brune T, Lindberg L, Waldenstrom U. The Stockholm Neonatal Family Centered Care Study: effects on length of stay and infant morbidity. Pediatrics. 2010 Feb;125(2):e278-85. doi: 10.1542/peds.2009-1511. Epub 2010 Jan 25. PMID 20100748
- [Background] Palisano R, Rosenbaum P, Walter S, Russell D, Wood E, Galuppi B. Development and reliability of a system to classify gross motor function in children with cerebral palsy. Dev Med Child Neurol. 1997 Apr;39(4):214-23. doi: 10.1111/j.1469-8749.1997.tb07414.x. PMID 9183258
- [Background] Pineda RG, Neil J, Dierker D, Smyser CD, Wallendorf M, Kidokoro H, Reynolds LC, Walker S, Rogers C, Mathur AM, Van Essen DC, Inder T. Alterations in brain structure and neurodevelopmental outcome in preterm infants hospitalized in different neonatal intensive care unit environments. J Pediatr. 2014 Jan;164(1):52-60.e2. doi: 10.1016/j.jpeds.2013.08.047. Epub 2013 Oct 17. PMID 24139564
- [Background] Wood-Kaczmar A, Deas E, Wood NW, Abramov AY. The role of the mitochondrial NCX in the mechanism of neurodegeneration in Parkinson's disease. Adv Exp Med Biol. 2013;961:241-9. doi: 10.1007/978-1-4614-4756-6_20. PMID 23224884
- [Background] Vohr B, McGowan E, McKinley L, Tucker R, Keszler L, Alksninis B. Differential Effects of the Single-Family Room Neonatal Intensive Care Unit on 18- to 24-Month Bayley Scores of Preterm Infants. J Pediatr. 2017 Jun;185:42-48.e1. doi: 10.1016/j.jpeds.2017.01.056. Epub 2017 Feb 24. PMID 28238479
- [Background] White RD, Smith JA, Shepley MM; Committee to Establish Recommended Standards for Newborn ICU Design. Recommended standards for newborn ICU design, eighth edition. J Perinatol. 2013 Apr;33 Suppl 1:S2-16. doi: 10.1038/jp.2013.10. PMID 23536026
- [Background] Bayley, N. (2006). Bayley Scales of Infant and Toddler Development: Technical manual (3rd ed.). San Antonio, TX: Harcourt Assessment, Inc.
- [Background] Stevens, D. C., Munson, D. P., & Khan, M. A. (2016). The single-family room neonatal intensive care environment. NeoReviews, 17(12)(17(12)), e687-e696.
- See also: Winnipeg Regional Health Authority. Winnipeg Assessment of Neonatal Nurses Need Tool (WANNNT). Retrieved 01/15, 2018 — http://cna-aiic.ca/~/media/cna/files/safe-staffing-toolkit/WANNNT-2013.pdf

DOCUMENTS (2):
  • Informed Consent Form (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT03867669/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03867669/Prot_SAP_001.pdf